CLINICAL TRIAL: NCT00922259
Title: Phase 1 Inpatient Study of the Safety and Immunogenicity of Live Influenza A Vaccine H7N7 (6-2) AA ca Recombinant (A/Netherlands/219/03 (H7N7) x A/Ann Arbor/ 6/60 ca), a Live Attenuated Virus Vaccine Candidate for Prevention of Avian Influenza H7N7 Infection in the Event of a Pandemic
Brief Title: Safety and Immunogenicity of Live Influenza A Vaccine for Avian Influenza H7N7
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: URMC 10-003
Record Dates: First submitted 2009-05-28; First posted 2009-06-17 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Influenza A
Keywords: Flu; Influenza; Vaccine; Prevention
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- H7N7 Vaccine (Experimental): Participants will be administered two doses of the candidate live influenza A H7N7 vaccine
  Interventions: Biological: Influenza A H7N7 vaccine

INTERVENTIONS:
Biological: Influenza A H7N7 vaccine — Participants will be administered two doses of the candidate vaccine at a dosage of approximately 10^7.5 50% tissue culture infectious dose (TCID50), in the form of nasal spray. The doses will be administered 28-62 days apart.

SUMMARY:
Every year the human population suffers from seasonal outbreaks of influenza resulting in both illness and death. However, the rates of illness and death from seasonal outbreaks are significantly lower than those suffered during times of influenza pandemic, such as those experienced in 1918, 1957, and 1968. The reason for this difference lies in presence of immunity within a population. With seasonal outbreaks of influenza most people have some immunity to the circulating strain and usually only those with weakened immune systems experience serious complications. Influenza pandemics, in contrast, are the result of a completely new viral subtype to which nobody possesses an immunity, leaving everyone vulnerable to the most serious of complications.

It has been estimated that the next flu pandemic could cause over 200,000 deaths and over 700,000 hospitalizations in the US alone. The need for an effective viral vaccine is high. The purpose of this study is to test the safety and immunogenicity of a live influenza A strain vaccine, which would be able to combat an influenza pandemic.

DETAILED DESCRIPTION:
Influenza, also called the flu, is an RNA virus belonging to the family Orthomyxoviridae that consists of 4 genera: influenza A, influenza B, influenza C, and Thogoto viruses. This vaccine study focuses on influenza A. Influenza A viruses are widely distributed in nature and can infect a wide variety of birds and mammals, including humans. Influenza viral infections affect the respiratory system and are particularly dangerous for those with weakened immune systems.

Within the influenza A genus, there are several viral subtypes classified by the ability to produce an immune response of their surface glycoproteins, hemagglutinin (HA) and neuraminidase (NA). In contrast to other species, influenza A has relatively few subtypes capable of triggering outbreaks within the human population. Only viruses bearing both H1, H2, or H3 HA genes, and N1 or N2 NA genes have circulated among the human population throughout the 20th century. The years 1918, 1957, and 1968 were all marked by extremely high rates of morbidity and mortality related to influenza. These were also the years in which novel subtypes of influenza had begun to circulate among the population. Because the human immune system had not yet created antibodies for these viruses, the population easily succumbed to a flu outbreak which consequently left thousands dead or impaired. It has been estimated that the next flu pandemic could cause upwards of 200,000 deaths and possibly over 700,000 hospitalizations.

Transmission of influenza subtypes through waterfowl, known as avian influenzas (AI), is of particularly great concern to the human population because it has the potential to cause a human influenza pandemic. In the last decade, it has been the AI viruses which have claimed the lives of hundreds during outbreaks.

At the start of a pandemic, all humans are immunologically naïve if the nascent virus contains antigenically novel HA and NA subtypes. In the event of a pandemic, the need for an effective vaccine is unequivocal. This study will test the safety, infectivity, and immunogenicity of a live-attenuated pandemic virus vaccine. The study will be an open-label, inpatient trial that will be initiated between April 1st and December 20th of each calendar year, when wild-type influenza virus is unlikely to be circulating in the community. Eligible participants will attend a study screening, which includes medical history, physical examination, hematology testing, liver and renal function testing, H7N7 antibody titer, HIV and Hepatitis B and C screening, urine dipstick testing (with possible urinalysis in the event of an abnormal urine dipstick result), and urine drug toxicology testing. Female participants of child-bearing age may also have a pregnancy test.

Two days prior to each vaccination, participants will be admitted to the isolation unit in order to become familiar with unit procedures. There will be two vaccinations during the course of the study. On the day of the first vaccination, a physical examination will be performed and all female participants will have a urine pregnancy test. Only if the participant is deemed healthy will a dose of vaccine in the form of nasal spray will be administered.

Following vaccination, all participants will remain on the isolation unit for at least 9 days. Physical examination and test of NW for influenza virus culture will be performed daily until discharge. They will be discharged once nasal wash (NW) specimens test negative for influenza for at least 2 consecutive days beginning on or after Day 7. Physical examination and NW for influenza virus culture will be performed daily until discharge. Participants will return for inpatient treatment 26 days after receiving their first dose of the vaccine. Two days later, or 28 days after the first vaccine, participants will receive a second dose of the influenza vaccine. Participants will then follow the same procedures as before, undergoing daily physical exams and testing of NW specimens. They will be eligible for discharge after another 9 days, provided their NW specimens test negative for influenza for 2 consecutive days.

All participants will undergo follow-up testing 56, 82, and 208 days after receiving the first dose of the vaccine. This testing will include providing an interim history, assessment for severe adverse events (SAEs), collection of a blood sample, completing a nasal wash, and assessment for treatments that could potentially interfere with vaccine-induced immunity.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* General good health, without significant medical illness, physical examination findings, or significant laboratory abnormalities as determined by the investigator
* Available for the duration of the trial
* Female participants must agree to use effective birth control methods for the duration of the study. More information on this criterion can be found in the study protocol.
* Agrees to store blood specimens for future research

Exclusion Criteria:

* Pregnancy or breast-feeding
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies including urine testing. Clinically significant ALT levels, as determined by the Principal Investigator, will be exclusionary at baseline, prior to vaccination.
* Behavioral or cognitive impairment or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the study protocol
* Previous enrollment in an H7 influenza vaccine trial or in any study of an avian influenza vaccine
* Seropositive to the H7N7 influenza A virus (serum HI titer greater than 1:8)
* Positive urine drug toxicology test indicating narcotic use or dependency
* Have medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant participating in the trial or would render the participant unable to comply with the protocol
* History of anaphylaxis
* Allergy to oseltamivir
* Diagnosis of asthma or reactive airway disease within the past 2 years
* History of Guillain-Barre Syndrome
* Positive ELISA and confirmatory Western blot tests for HIV-1
* Positive ELISA and confirmatory test (for example, recombinant immunoblot assay [RIBA]) for hepatitis C virus (HCV)
* Positive test for hepatitis B virus surface antigen (HBsAg) by ELISA.
* Known immunodeficiency syndrome
* Use of corticosteroids (excluding topical preparations) or immunosuppressive drugs within 30 days prior to vaccination
* Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to study vaccination
* History of a surgical splenectomy
* Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to study vaccination
* Current smoker unwilling to stop smoking for the duration of the study. More information on this criterion can be found in the study protocol.
* Travel to the Southern Hemisphere within 14 days prior to study vaccination.
* Travel on a cruise ship within 14 days prior to study vaccination
* Current involvement with the poultry industry. This refers to direct contact with poultry within the 14 days prior to the study or after the study completion.
* Receipt of another investigational vaccine or drug within 30 days prior to study vaccination
* Allergy to eggs or egg products

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2010-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Immunogenicity as measured by Anti-H7N7 antibody and seroconversion | Measured on Days 2 to 9 and 26 to 37
Determine the frequency of vaccine-related reactogenicity events (REs) and other adverse events (AEs) for 2 doses of vaccine | Measured on Days 2 to 9 and 26 to 37

SECONDARY OUTCOMES:
Frequency of vaccine-related reactogenicity events (REs) and other adverse events (AEs) for each dose | Measured on Days 2 to 9 and 26 to 37
Area under the curve of nasal virus shedding after each dose of vaccine | Measured on Days 2 to 9 and 28 to 37
Amount of serum and nasal wash antibody induced by the vaccine | Measured through Day 208
Number of vaccinees infected with the H7N7 NL 2003/AA ca recombinant vaccine candidate | Measured through Day 208
Phenotypic stability of vaccine virus shed | Measured through Day 208
Determination of whether immunogenicity is enhanced by a second dose of vaccine, and whether the first dose of vaccine restricts replication of the second dose | Measured through Day 208
T-cell mediated and innate immune responses against the H7N7 NL 2003/AA ca recombinant vaccine candidate | Measured through Day 208
Development of serum antibody, as assessed by either hemagluttinin (HAI) or microneutralization (MN) assays | Measured through Day 208

CONTACTS AND LOCATIONS:
Overall Officials: John Treanor, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Background] Kelly H, Carville K, Grant K, Jacoby P, Tran T, Barr I. Estimation of influenza vaccine effectiveness from routine surveillance data. PLoS One. 2009;4(3):e5079. doi: 10.1371/journal.pone.0005079. Epub 2009 Mar 31. PMID 19333374
- [Background] Roose K, Fiers W, Saelens X. Pandemic preparedness: toward a universal influenza vaccine. Drug News Perspect. 2009 Mar;22(2):80-92. doi: 10.1358/dnp.2009.22.2.1334451. PMID 19330167
- [Background] Schwehm M, Wilson N. Potential impact of pandemic influenza interventions in New Zealand: a brief modelling study. N Z Med J. 2009 Mar 13;122(1291):117-21. No abstract available. PMID 19322265